CLINICAL TRIAL: NCT00944281
Title: A Randomized, Double-blind, Controlled Trial in Rural Burkina Faso to Determine the Optimal Amount of Zinc to Include in a Lipid-based Nutrient Supplement (LNS). Part of the iLiNS Study
Brief Title: Optimal Amount of Zinc to Include in a Lipid-based Nutrient Supplement (LNS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Université Polytechnique de Bobo-Dioulasso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 236850; iLiNS-Zinc
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Malnutrition
Keywords: point-of-use fortification; zinc supplement; lipid-based nutrient supplement; zinc deficiency; micronutrient deficiency; anemia
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- LNS-Zn5 (Experimental): Daily intake of 20 g LNS containing 5 mg of zinc and a daily placebo supplement
  Interventions: Dietary Supplement: LNS-Zn5
- LNS-Zn10 (Experimental): Daily intake of 20 g LNS containing 10 mg of zinc and a daily placebo supplement
  Interventions: Dietary Supplement: LNS-Zn10
- LNS-Zn0 (Placebo Comparator): Daily intake of 20 g LNS containing 0 mg of zinc and a daily placebo supplement
  Interventions: Dietary Supplement: LNS-Zn0
- Suppl-Zn5 (Experimental): Daily intake of zinc supplement containing 5 mg of zinc and 20 g LNS containing 0 mg of zinc
  Interventions: Dietary Supplement: Suppl-Zn5
- Delayed intervention group (No Intervention): Standard care from age 8 to 18 months. Daily consumption of LNS from age 18 to 28 months.

INTERVENTIONS:
Dietary Supplement: LNS-Zn5 — Daily consumption of 20 g LNS containing 5 mg of zinc and daily placebo supplement
  Other Names: Nutriset
  Arms: LNS-Zn5
Dietary Supplement: LNS-Zn10 — Daily consumption of 20 g LNS containing 10 mg of zinc and daily placebo supplement
  Other Names: Nutriset
  Arms: LNS-Zn10
Dietary Supplement: LNS-Zn0 — 20 g of LNS containing 0 mg of zinc and a daily placebo supplement
  Other Names: Nutriset
  Arms: LNS-Zn0
Dietary Supplement: Suppl-Zn5 — Daily 5 mg zinc supplement ant consumption of 20 g LNS containing 0 mg of zinc
  Other Names: Nutriset
  Arms: Suppl-Zn5

SUMMARY:
To assess zinc-related biochemical and functional responses among young Burkinabe children with a presumed high risk of zinc deficiency who receive micronutrient products containing different amounts of zinc, provided with or between meals.

DETAILED DESCRIPTION:
Young healthy children will be identified by periodic consensus in the study area. 3200 infants meeting a set of eligibility criteria will be randomly assigned to receive lipid-based nutrient supplements (LNS) with different amounts of zinc and a placebo or zinc supplement from 9 to 18 months of age. The families will receive the respective supplement at weekly intervals and the participants undergo a morbidity evaluation weekly, anthropometric evaluation at 9, 12, 15 and 18 months and laboratory analyses at enrollment and at 18 months of age. Growth outcomes will be analyzed during the two-year follow up at 24, 30, 36 and 42 months of age.

ELIGIBILITY:
Inclusion Criteria:

* 9.0 to 9.9 mo of age

Exclusion Criteria:

* severe anemia
* severely malnourished
* presence of bipedal oedema
* severe illness
* congenital abnormalities
* chronic medical condition
* known HIV infection of mother or infant
* history of peanut allergy
* history of anaphylaxis or serious allergic reaction to any substance

Ages: 9 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3220 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in length and length-for-age Z-score | 9 to 18 mo of age
Change in weight and weight-for-age Z-score | 9 to 18 mo of age
Incidence of diarrhea and laboratory-confirmed malaria infection | 9 to 18 mo of age
Change in plasma zinc concentration | 9 to 18 mo of age
Change in body composition | 9 to 18 mo of age

SECONDARY OUTCOMES:
Change in head circumference and mid-upper arm circumference | 9 to 18 mo of age
Change in stunting, underweight, and wasting | 9 to 18 mo of age
Change in hemoglobin, iron, vitamin A and iodine status | 9 to 18 mo of age
Incidence of acute lower respiratory infection (ALRI) | 9 to 18 mo of age

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Dewey, PhD, Study Director — University of California, Davis; Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Institut de Recherche en Sciences de la Sante, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Result] Hess SY, Abbeddou S, Jimenez EY, Some JW, Vosti SA, Ouedraogo ZP, Guissou RM, Ouedraogo JB, Brown KH. Small-quantity lipid-based nutrient supplements, regardless of their zinc content, increase growth and reduce the prevalence of stunting and wasting in young burkinabe children: a cluster-randomized trial. PLoS One. 2015 Mar 27;10(3):e0122242. doi: 10.1371/journal.pone.0122242. eCollection 2015. PMID 25816354
- [Result] Some JW, Abbeddou S, Yakes Jimenez E, Hess SY, Ouedraogo ZP, Guissou RM, Vosti SA, Ouedraogo JB, Brown KH. Effect of zinc added to a daily small-quantity lipid-based nutrient supplement on diarrhoea, malaria, fever and respiratory infections in young children in rural Burkina Faso: a cluster-randomised trial. BMJ Open. 2015 Sep 11;5(9):e007828. doi: 10.1136/bmjopen-2015-007828. PMID 26362661
- [Result] Hess SY, Abbeddou S, Yakes Jimenez E, Ouedraogo JB, Brown KH. Iodine status of young Burkinabe children receiving small-quantity lipid-based nutrient supplements and iodised salt: a cluster-randomised trial. Br J Nutr. 2015 Dec 14;114(11):1829-37. doi: 10.1017/S0007114515003554. Epub 2015 Sep 28. PMID 26411504
- [Result] Abbeddou S, Yakes Jimenez E, Some JW, Ouedraogo JB, Brown KH, Hess SY. Small-quantity lipid-based nutrient supplements containing different amounts of zinc along with diarrhea and malaria treatment increase iron and vitamin A status and reduce anemia prevalence, but do not affect zinc status in young Burkinabe children: a cluster-randomized trial. BMC Pediatr. 2017 Feb 2;17(1):46. doi: 10.1186/s12887-016-0765-9. PMID 28152989
- [Result] Hess SY, Peerson JM, Becquey E, Abbeddou S, Ouedraogo CT, Some JW, Yakes Jimenez E, Ouedraogo JB, Vosti SA, Rouamba N, Brown KH. Differing growth responses to nutritional supplements in neighboring health districts of Burkina Faso are likely due to benefits of small-quantity lipid-based nutrient supplements (LNS). PLoS One. 2017 Aug 3;12(8):e0181770. doi: 10.1371/journal.pone.0181770. eCollection 2017. PMID 28771493
- [Result] Abbeddou S, Hess SY, Yakes Jimenez E, Some JW, Vosti SA, Guissou RM, Ouedraogo JB, Brown KH. Comparison of methods to assess adherence to small-quantity lipid-based nutrient supplements (SQ-LNS) and dispersible tablets among young Burkinabe children participating in a community-based intervention trial. Matern Child Nutr. 2015 Dec;11 Suppl 4(Suppl 4):90-104. doi: 10.1111/mcn.12162. PMID 25521188
- [Derived] Abbeddou S, Jimenez EY, Hess SY, Some JW, Ouedraogo JB, Brown KH. Small-quantity lipid-based nutrient supplements, with or without added zinc, do not cause excessive fat deposition in Burkinabe children: results from a cluster-randomized community trial. Eur J Nutr. 2022 Dec;61(8):4107-4120. doi: 10.1007/s00394-022-02936-6. Epub 2022 Jul 13. PMID 35829783
- [Derived] Prado EL, Abbeddou S, Adu-Afarwuah S, Arimond M, Ashorn P, Ashorn U, Brown KH, Hess SY, Lartey A, Maleta K, Ocansey E, Ouedraogo JB, Phuka J, Some JW, Vosti SA, Yakes Jimenez E, Dewey KG. Linear Growth and Child Development in Burkina Faso, Ghana, and Malawi. Pediatrics. 2016 Aug;138(2):e20154698. doi: 10.1542/peds.2015-4698. PMID 27474016
- [Derived] Prado EL, Abbeddou S, Yakes Jimenez E, Some JW, Ouedraogo ZP, Vosti SA, Dewey KG, Brown KH, Hess SY, Ouedraogo JB. Lipid-Based Nutrient Supplements Plus Malaria and Diarrhea Treatment Increase Infant Development Scores in a Cluster-Randomized Trial in Burkina Faso. J Nutr. 2015 Apr 1;146(4):814-822. doi: 10.3945/jn.115.225524. PMID 26962193
- See also: PLoS ONE: Small-quantity lipid-based nutrient supplements... — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0122242